CLINICAL TRIAL: NCT06734754
Title: The Effect of Fetal Heart Sound Played by Parents Diagnosed With Risky Pregnancy on Attachment and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hilal Dincer, Inonu University, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Inonu U.
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Attachment; Risk Pregnancy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): fetal heart sound listening
  Interventions: Device: fetal heart sound listening
- Control Group (No Intervention): fetal heart sound was not played

INTERVENTIONS:
Device: fetal heart sound listening — The pregnant women in the experimental group and their partners listened to fetal heart sounds for 7 days. After obtaining pre-test data from the participants in the intervention group, the midwifery intervention to be implemented was explained. A fetal heart rate monitoring device, which will be given to couples to listen to the fetal heart sound before sleep, was introduced. They were told that they had to listen to the fetal heart sound at least 7 times using this device. A supporting application was downloaded to the pregnant woman's phone for the installation of the fetal heart rate monitoring device. The way of using the application and the operation steps were introduced. It was explained to the couples that the application can detect the baby's heartbeat within seconds thanks to its smart search technology, and also provides step-by-step guidance by giving live feedback.
  Arms: Experimental Group

SUMMARY:
The research was designed as a randomized controlled experimental type to determine the effect of fetal heart sound played to parents diagnosed with risky pregnancies on attachment and anxiety. With the results obtained from this study, it is aimed to contribute to the limited literature on the effect of fetal heart sound played to parents diagnosed with risky pregnancy on attachment and anxiety.

Research question or Hypothesis(ies) and Purpose(s):

The purpose of this study is to determine the effect of fetal heart sound played to parents diagnosed with high-risk pregnancy on attachment and anxiety.

H1-a: Listening to the fetal heart sound reduces the anxiety level of the expectant mother.

H1-b: Listening to the fetal heart sound increases the maternal attachment of the expectant mother.

H1-c: Listening to the fetal heart sound reduces the anxiety level of the expectant father.

H1-d: Listening to the fetal heart sound increases the paternal attachment of the expectant father.

The research will be conducted on 2 groups: 1 experimental and 1 control group. In order to obtain pre-test data of the research, couples will fill in the determined measurement tools. The couples' contact information will be recorded, their appointment dates will be determined and an appointment card will be issued. The intervention applied by the researcher to the participants in the experimental group will be completed in 7 days. At the end of the 7th day, post-test data will be obtained using measurement tools.

Pretest data will be obtained using measurement tools in the first interview with the control group. No interventional intervention will be applied to the participants in the control group by the researcher. Post-test data will be obtained 7 days later by applying the same measurement tools.

DETAILED DESCRIPTION:
Criteria for Inclusion in the Research:

* Being diagnosed with a risky pregnancy (pregnancy under 18 years of age, pregnancy over 35 years of age, birth interval of less than two years, experiencing one of the prenatal hemorrhages, premature rupture of membranes, hypertensive conditions during pregnancy, hyperemesis gravidarum, multiple pregnancies, gestational diabetes, placenta previa , having a medical disease history such as polyhydramnios, oligohydramnios, heart disease, thyroid diseases, blood diseases, experiencing one of the infectious diseases, Rh incompatibility, getting pregnant with assisted reproductive techniques, varicose veins, smoking, alcohol, substance use)
* No verbal communication or reading and writing disabilities,
* Has a smart phone and internet access,
* 27-38. week of pregnancy,
* Women who agreed to participate in the study voluntarily and whose consent was obtained
* Pregnant women who were not previously or currently diagnosed with a psychiatric disease were included in the sample.

Criteria for Exclusion from the Research:

* Participating in the study and then deciding to leave,
* Those who fill out the data forms incompletely or do not complete them will be excluded from the research.Exclusion Criteria from the Study:
* Not diagnosed with high-risk pregnancy,
* Those who do not live with their spouse,
* Unmarried
* Pregnant women with communication difficulties or mental disabilities were not included in the study.

Variables of the research:

Independent Variable of the Research: Demographic characteristics of the couples Dependent Variable of the Research: Couples' attachment and anxiety states Control variables of the study: Some individual characteristics of the couples (age, education, income level, employment status, place of residence)

Data collection tools:

While data were being collected, Personal Information Form-Female , Personal Information Form-Male , "Prenatal Mother Attachment Scale ", "Prenatal Father Attachment Scale " and "State Anxiety Scale" were used ".

ELIGIBILITY:
Inclusion Criteria:

* • Being diagnosed with a risky pregnancy (pregnancy under 18 years of age, pregnancy over 35 years of age, birth interval of less than two years, experiencing one of the prenatal hemorrhages, premature rupture of membranes, hypertensive conditions during pregnancy, hyperemesis gravidarum, multiple pregnancies, gestational diabetes, placenta previa Having a history of medical diseases such as polyhydramnios, oligohydramnios, heart disease, thyroid diseases, having blood diseases, infectious diseases, Rh incompatibility, pregnancy with assisted reproductive techniques, varicose veins, smoking, alcohol, substance use)

  * No verbal communication or reading and writing disabilities,
  * Having a smartphone and internet access,
  * 27-38. week of pregnancy,
  * Women who agreed to participate in the study voluntarily and whose consent was obtained
  * Pregnant women who were not previously or currently diagnosed with a psychiatric disease were included in the sample.

Exclusion Criteria:

* • Not diagnosed with high-risk pregnancy,

  * Those who do not live with their spouse,
  * Unmarried
  * Pregnant women with communication difficulties or mental disabilities were not included in the study.
  * Participating in the study and then deciding to leave,
  * Those who fill out the data forms incompletely or do not complete them will be excluded from the research.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 272 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The effect of auscultated fetal heart sound on the anxiety level of the expectant mother | 7 days
  State Anxiety Scale: It is scored according to the severity of the emotions or behaviors expressed in the scale as (1) not at all, (2) a little, (3) a lot, (4) completely. The 10 items of the scale are reverse scored: 1, 2, 5, 8, 10, 11, 15, 16, 19, 20. A score of 4 from the scale indicates high anxiety in plain expressions, while it indicates low anxiety in reverse expressions. When calculating the scale score, 50 points are added to the difference between the total weighted scores of reverse expressions and plain expressions, and the total score varies between 20-80. A score below 36 indicates no anxiety, a score between 37 and 42 indicates mild anxiety, and a score of 42 and above indicates high anxiety.
The effect of auscultated fetal heart sound on the maternal attachment of the expectant mother. | 7 days
  Prenatal Maternal Attachment Scale consists of 19 items and two subscales. The scale is a 5-point Likert type, 11 items are reverse scored and the items take values between 1-5. A high score from the scale indicates a high degree of attachment.
The effect of auscultated fetal heart sound on the anxiety level of the expectant father | 7 days
  State Anxiety Scale: It is scored according to the severity of the emotions or behaviors expressed in the scale as (1) not at all, (2) a little, (3) a lot, (4) completely. The 10 items of the scale are reverse scored: 1, 2, 5, 8, 10, 11, 15, 16, 19, 20. A score of 4 from the scale indicates high anxiety in plain expressions, while it indicates low anxiety in reverse expressions. When calculating the scale score, 50 points are added to the difference between the total weighted scores of reverse expressions and plain expressions, and the total score varies between 20-80. A score below 36 indicates no anxiety, a score between 37 and 42 indicates mild anxiety, and a score of 42 and above indicates high anxiety.
The effect of fetal heart sound playback on paternal attachment | 7 days
  Prenatal Father Attachment Scale consists of 16 items and two subscales. Increasing score indicates higher degree of attachment. The scale is a 5-point Likert type and 9 items are reverse scored.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal, Malatya, Yeşilyurt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No